CLINICAL TRIAL: NCT01426113
Title: A Study of the Safety and Efficacy of Bimatoprost Ophthalmic Solution in Paediatric Patients With Glaucoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to corporate decision.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-056
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bimatoprost ophthalmic solution formulation A and vehicle (Experimental): 1 drop bimatoprost vehicle in the affected eye(s) in the morning and 1 drop of bimatoprost ophthalmic solution formulation A in the affected eye(s) in the evening for 6 weeks, followed by 1 drop bimatoprost ophthalmic solution formulation A in the affected eye(s) in the morning and 1 drop bimatoprost vehicle in the affected eye(s) in the evening for 6 additional weeks.
  Interventions: Drug: bimatoprost ophthalmic solution formulation A; Drug: bimatoprost vehicle
- timolol ophthalmic solution (Active Comparator): 1 drop timolol ophthalmic solution in the affected eye(s) in the morning and evening for 12 weeks.
  Interventions: Drug: timolol ophthalmic solution

INTERVENTIONS:
Drug: bimatoprost ophthalmic solution formulation A — 1 drop of bimatoprost ophthalmic solution formulation A in the affected eye(s) in the evening for 6 weeks, followed by 1 drop of bimatoprost ophthalmic solution formulation A in the affected eye(s) in the morning for 6 weeks.
  Arms: bimatoprost ophthalmic solution formulation A and vehicle
Drug: timolol ophthalmic solution — 1 drop timolol ophthalmic solution in the affected eye(s) in the morning and evening for 12 weeks.
  Arms: timolol ophthalmic solution
Drug: bimatoprost vehicle — 1 drop of bimatoprost vehicle in the affected eye(s) in the morning for 6 weeks, followed by 1 drop of bimatoprost vehicle in the affected eye(s) in the evening for 6 weeks.
  Arms: bimatoprost ophthalmic solution formulation A and vehicle

SUMMARY:
The purpose of this study is to assess the safety and efficacy of a new formulation of bimatoprost ophthalmic solution compared to timolol ophthalmic solution in the treatment of paediatric patients with glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital, juvenile glaucoma
* Requires treatment with IOP-lowering medication in one or both eyes

Exclusion Criteria:

* Surgical intervention is indicated or planned to lower IOP
* Abnormally low body weight (below 5th percentile)
* Any active eye infection or disease
* Anticipated use of contact lenses during the study
* Topical ocular steroid use within 2 months
* History of ocular trauma in either eye
* Required chronic use of ocular medications (other than study medication) during the study (intermittent use of artificial tears permitted)

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (9):
- Louisville, Kentucky, United States
- Amiens, France
- Italy (2):
  - Milan
  - Parma
- Philippines (2):
  - City of Taguig
  - Makati
- Seoul, South Korea
- Taipei, Taiwan
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was discontinued prematurely after enrollment of 6 patients.
Period: Overall Study
Arm/Group | Bimatoprost Ophthalmic Solution Formulation A and Vehicle | Timolol Ophthalmic Solution
Started | 3 | 3
Completed | 2 | 1
Not Completed | 1 | 2
Not completed — Study Discontinued | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost Ophthalmic Solution Formulation A and Vehicle | Timolol Ophthalmic Solution | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Customized [Number; unit: Participants]
  12 to 15 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP) in the Study Eye
Description: IOP is a measure of the fluid pressure inside the study eye. A negative number change from baseline indicates a reduction in IOP (improvement) and a positive change from baseline indicates an increase in IOP (worsening). Due to lack of enrollment, analysis was not performed for this outcome measure.
Time Frame: Baseline, Week 6
Population: Due to early termination of the study, no statistical analysis was performed and no data summaries were generated. From a target of 120 patients, only 6 patients (3 in each group) were enrolled.
Arm/Group | Bimatoprost Ophthalmic Solution Formulation A and Vehicle | Timolol Ophthalmic Solution
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Bimatoprost Ophthalmic Solution Formulation A and Vehicle | Timolol Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Ophthalmic Solution Formulation A and Vehicle (N=3) | Timolol Ophthalmic Solution (N=3)
Eyelash Hyperpigmentation (Eye disorders) | 0 | 1
Growth of Eyelashes (Eye disorders) | 1 | 1
Intraocular Pressure Increased (Investigations) | 0 | 1
Conjunctival Hyperaemia (Eye disorders) | 2 | 0
Eyelid Oedema (Eye disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Blepharal Pigmentation (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.